CLINICAL TRIAL: NCT01139840
Title: Vitamin D Status: Relative Efficacy of Vitamins D2 and D3
Brief Title: Relative Efficacy of Vitamins D2 and D3 in Adult Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: Health Future Foundation (Unknown); BTR Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 09-15612
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: vitamin D2; vitamin D3; ergocalciferol; cholecalciferol; vitamin D status; To determine relative potency of vitamins D2 and D3 under conditions of continuous administration; To determine change in vitamin D content of subcutaneous fat after 12 weeks' administration
MeSH Terms: interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin D2 (Active Comparator)
  Interventions: Dietary Supplement: vitamin D2
- vitamin D3 (Active Comparator)
  Interventions: Dietary Supplement: vitamin D3

INTERVENTIONS:
Dietary Supplement: vitamin D2 — Study Supplement
  Arms: vitamin D2
Dietary Supplement: vitamin D3 — Study Supplement
  Arms: vitamin D3

SUMMARY:
Vitamin D2 in chronic dosing will produce less of an elevation of serum 25(OH)D than will the same dose of vitamin D3.

ELIGIBILITY:
Inclusion Criteria:

* willingness to withhold supplement use for duration of study
* willingness to avoid sun exposure for duration of study

Exclusion Criteria:

* vitamin D supplement use
* conditions that affect vitamin D metabolism by the body

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
AUC for increment in serum 25(OH)D | 12 weeks

SECONDARY OUTCOMES:
change in vitamin D content of subcutaneous fat | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Heaney, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Heaney RP, Recker RR, Grote J, Horst RL, Armas LA. Vitamin D(3) is more potent than vitamin D(2) in humans. J Clin Endocrinol Metab. 2011 Mar;96(3):E447-52. doi: 10.1210/jc.2010-2230. Epub 2010 Dec 22. PMID 21177785